CLINICAL TRIAL: NCT01577108
Title: Oral Probiotics Lactobacillus Rhamnosus GR-1 and Lactobacillus Reuteri RC-14 Reduce Group B Streptococci Colonization in Pregnant Women
Brief Title: Oral Probiotics Reduce Group B Streptococci Colonization in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: DMR99-IRB-309
Record Dates: First submitted 2011-07-20; First posted 2012-04-13 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-02

CONDITIONS: Group B Streptococcal Infection
Keywords: 31-32 Weeks of Gestation Completed; Group B Streptococcal Infection; Streptococcus Group B Infection of the Infant
MeSH Terms: conditions — Streptococcal Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotics, GBS Test (Experimental): Treated with 2 oral probiotics once daily before sleeping for 14 days
  Interventions: Dietary Supplement: Probiotic
- Non-probiotics, GBS test (Placebo Comparator): Treated with 2 placebo capsules once daily before sleeping for 14 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — oral taking 2 capsules before sleeping per day for 14 days
  Other Names: U-relax oral capsule, Lactobacillus GR-1 and RC-14
  Arms: Probiotics, GBS Test
Dietary Supplement: Placebo — oral taking 2 capsules before sleeping per day for 14 days
  Other Names: Placebo oral capsule
  Arms: Non-probiotics, GBS test

SUMMARY:
The purpose of this study is to examine whether daily use of oral gelatin capsules containing dried viable Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14 can reduce the GBS colonization rate of vagina and rectum in pregnant women who present with GBS-positive diagnosed by GBS culture at 35-37 weeks gestation.

This study is a prospective double blind randomized clinical trial. Vaginal and rectal GBS screening culture are carried out for all pregnant women at 35-37 weeks of gestation in our out-patient department. Subjects with vagina and rectum GBS colonization are invited to participate in our study after informed consent. A total of 200 pregnant women will participate in the study during the 12-months trial period. They are randomly assigned to one of the two groups. The study group is treated with two oral capsules of probiotics once daily (before sleeping) for 14 days, and the control group will take 2 capsules of placebos. Vaginal and rectal GBS culture is repeated for all participators 2 weeks later. All participators will treated according to GBS guideline by CDC in 2002 during laboring.

DETAILED DESCRIPTION:
Group B streptococci (GBS) colonizes the vagina and rectum in 10-30% of pregnant women. In the newborn, GBS is a leading cause of neonatal sepsis and a major cause of pneumonia and meningitis. Intrapartum penicillin G prophylaxis aims to prevent early-onset group B streptococci (GBS) sepsis by interrupting vertical transmission. According to the Center of Disease Control and Prevention (CDC) guideline in 2002, a minimum of 4 hours of intrapartum antibiotics prophylaxis is generally recommended to prevent early-onset group B Streptococcous (GBS) because less than 4 hours may not achieve adequate levels drugs. Even with the most valiant of efforts, there will frequently be GBS-positive mothers who arrive at the labor floor and deliver in fewer than 4 hours, especially in multiparous mothers. Preliminary studies as well as data from a large health maintenance organization demonstrated the 40-50%of GBS-colonized women do not receive antibiotics at least 4 hours before delivery due the rapidity of their labors. Newborns of all GBS-positive women who present to labor units and deliver before receiving 4 hours of intrapartum antibiotic prophylaxis are deemed as "at risk" and recommended to undergo blood cultures, complete blood count, and 48 hours of observation. This problem is not easily resolved by antibiotic treatment of the pathogen; thus, such tranditional approaches to patient management need to be re-evaluated.

Probiotics are defined as live micro-organisms which, when administered in an adequate amount, confer a health benefit on the host. Probiotics have been shown to displace and kill pathogens and modulate the immune response by interfering with the inflammatory cascade that leads to preterm labour and delivery. Lactobacilli are the dominant bacteria of vaginal flora and possess antimicrobial properties that regulate other urogenital microbiota. Incomplete cure and recurrence of genitourinary infections lead to a shift of the local flora from a predominance of lactobacilli to coliform uropathogens. Use of Lactobacillus-containing probiotics to restore commensal vaginal flora has been proposed for the treatment and prophylaxis of bacterial urogenital infections. The actual mechanism of action of probiotics in the vagina is probably multifactorial. The production of lactic acid, bacteriocin, and hydrogen peroxide seems to be important, and modulation of immunity is another possible mechanism. The administration of these Lactobacilli by mouth or intravaginally, or both has been shown to be safe and effective in reducing, or treating, or both, urogenital infections. For pregnant women, such restoration could be important to prevent BV and lower the risk of PTL Daily use of oral gelatin capsules containing dried viable Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14 has been shown to decreased e risk of bacterial vaginosis and maintain normal lactobacilli vaginal flora. These organisms are antagonistic to the growth and adhesion of various intestinal and urogenital pathogens including Salmonella typhimurium, Shigella sonnei, E coli 0157, toxic shock Staphylococcus aureus, group B streptococci, Enterococcus faecalis, G vaginalis, and uropathogenic E coli. In animal studies, these strains were found to be safe during pregnancy and to enhance the health of mothers and newborns. Studies are under way in Toronto, Ont, to test the effects of these strains on bacterial vaginosis in pregnant women at risk of preterm labour. These lactobacilli might also have a role in preventing vaginal colonization by group B streptococci, organisms that can cause serious illness and even death in newborns. Certain lactobacilli can inhibit growth and adhesion of streptococci in vitro, but whether they can do this in vivo is untested.

This study is a prospective double blind randomized clinical trial. Vaginal and rectal GBS screening culture are carried out for all pregnant women at 35-37 weeks of gestation in our OPD. Subjects with vagina and rectum GBS colonization are invited to participate in our study after informed consent. A total of 200 pregnant women will participate in the study during the 12-months trial period. They are randomly assigned to one of the two groups. The study group is treated with two oral capsules of probiotics once daily (before sleeping) for 14 days, and the control group will take 2 capsules of placebos. Vaginal and rectal GBS culture is repeated for all participators 2 weeks later. All participators will treated according to GBS guideline by CDC in 2002 during laboring.

Much of the current literature has investigated the potential of probiotics in preventing of bacterial vaginosis and preterm labor, but the usefulness of using probiotics as a surrogate or adjunctive therapy for intra-partum antibiotics prophylaxis in GBS colonized pregnant women dose not have any. This is the first study to investigate the role of probiotics in preventing and treating vaginal colonization by GBS in pregnant women. The purpose of this study is to examine whether oral taking Latobacillus-containing probiotics can reduce the GBS colonization rate of vagina and rectum in pregnant women who present with GBS-positive. Through the results of our study, we try to investigate the role of probiotics in preventing the unnecessary tests, admission and antibiotic treatment in newborn with GBS-positive mother who deliver fewer than 4 hours after laboring. We hope our results may have some effects on GBS sepsis protocols.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with positive GBS screening culture at 35-37 weeks of gestation
* singleton gestation
* subjects with agreement to abstain from the use of any systemic or intravaginal antibiotic, anti-fungal agents, or any other intravaginal product (i.e., contraceptive creams, gels, foams, sponges, lubricants, douches, etc) throughout the trial period

Exclusion Criteria:

* multiple gestations
* subjects with impaired immunity , diabetes or other significant disease or acute illness that in the investigator's assessment could complicate the evaluation
* vaginal or systemic antibiotics or antifungal therapy within 2 weeks of the screening visit.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ming Ho, MD, Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Probiotics, GBS Test: Treated with 2 oral probiotics once daily before sleeping for 14 days
  GR-1, RC-14: oral taking 2 capsules before sleeping per day for 14 days
- Non-probiotics, GBS Test: Treated with 2 placebo capsules once daily before sleeping for 14 days
  GR-1, RC-14: oral taking 2 capsules before sleeping per day for 14 days
Period: Overall Study
Arm/Group | Probiotics, GBS Test | Non-probiotics, GBS Test
Started | 54 | 56
Completed | 49 | 50
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotics, GBS Test | Non-probiotics, GBS Test | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 50 | 99
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 50 | 99
  Male | 0 | 0 | 0
Pregnancy, 35-37 weeks [Number; unit: Participants] | 49 | 50 | 99

OUTCOME MEASURES:

1. Primary Outcome: Number of GBS-Positive Pregnant Women Who Became GBS-Negative at Childbirth
Description: To exam the GBS colonization in both vagina and rectum when childbirth. The purpose of this study is to examine whether oral taking Lactobacillus-containing probiotics can reduce the GBS colonization rate of vagina and rectum in pregnant women who present with GBS-positive.
Time Frame: 2 weeks after taking probiotic
Population: The GBS colonization results changed from positive to negative in 21 women in the probiotic group (42.9%) and in nine women in the placebo group (18.0%) during this period.
Measure: Count of Participants; unit: Participants
Groups:
- Probiotics, GBS Test: Treated with 2 oral probiotics once daily before sleeping for 14 days
  GR-1, RC-14: oral taking 2 capsules before sleeping per day for 14 days
  Number of GBS-Positive pregnant women who became GBS-Negative at childbirth is 21 in the probiotic group (42.9%).
- Non-probiotics, GBS Test: Treated with 2 placebo capsules once daily before sleeping for 14 days
  GR-1, RC-14: oral taking 2 capsules before sleeping per day for 14 days
  Number of GBS-Positive pregnant women who became GBS-Negative at childbirth is 9 in the probiotic group (18.0%).
Arm/Group | Probiotics, GBS Test | Non-probiotics, GBS Test
Number analyzed (Participants) | 49 | 50
Participants | 21 | 9

ADVERSE EVENTS:
Time Frame: 2 to 4 weeks when taking probiotic capsules or placebo capsules
Arm/Group | Probiotics, GBS Test | Non-probiotics, GBS Test
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No